CLINICAL TRIAL: NCT06455033
Title: Effect of Manual Diaphragm Release Technique on Stepping Reaction Time and Balance in Patients with Chronic Obstructive Pulmonary Disease
Brief Title: Manual Diaphragm Release on Stepping Reaction Time in Chronic Obstructive Pulmonary Disease
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Beni-Suef University (Other)
Responsible Party: Principal Investigator, Mohammed Youssef Elhamrawy, Lecturer of Physical therapy, Beni-Suef University
Allocation: Non-Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: Manual Diaphragm Release
Record Dates: First submitted 2024-06-07; First posted 2024-06-12 (Actual); Last update posted 2024-10-15 (Actual); Status verified 2024-06

CONDITIONS: Respiratory Disease
MeSH Terms: conditions — Respiration Disorders | interventions — Breathing Exercises

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Study Group (Active Comparator): 30 patients with chronic obstructive pulmonary disease
  Interventions: Other: Manual Diaphragm Release Technique; Other: Breathing Exercise
- Control group (Active Comparator): 30 patients with chronic obstructive pulmonary disease
  Interventions: Other: Breathing Exercise

INTERVENTIONS:
Other: Manual Diaphragm Release Technique — The participant will assume a supine position with relaxed limbs. The therapist should position themselves at the head of the participant and make manual contact with the pisiform, hypothenar region, and the last three fingers on both sides, underneath the seventh to tenth rib costal cartilages. The therapist's forearms should be aligned towards the participant's shoulders. During the inspiratory phase, the therapist gently pulled the points of contact with both hands in the direction of the head and slightly laterally, accompanying the elevation of the ribs. During exhalation, the therapist deepens their contact towards the inner costal margin while maintaining resistance. As the respiratory cycles continues, the therapist progressively increases the depth of their contact within the costal margin.
  Arms: Study Group
Other: Breathing Exercise — Sit up straight in a chair lengthen the distance between your navel and sternum. Keep your shoulders relax.
  Keep the pelvis in neutral position (Sit on your sitting bones). Place your hands at either side of your lower ribs. Breath in slowly through your nose. As you inhale feel your ribs expanding outwards and upwards. During inhalation is generated expansion of the trunk in three directions front , sides and back.
  Breath out from your nose. As you exhale feel your lower ribs moving inwards.

SUMMARY:
Finding the effect of diaphragm release exercises on stepping reaction time and balance in patients with chronic obstructive pulmonary disease patients.

DETAILED DESCRIPTION:
Sixty patients with Chronic Obstructive Pulmonary Disease (COPD) will be randomly assigned to the experimental (EX) group and the control group (CON). The participants' age will be 55 years and above with history of COPD. The Ex group will attend 4 sessions/week of Manual Diaphragm Release Technique Combined with Deep Breathing (10:15-min) for 8 weeks, the CON will attend 4 sessions/week of Deep Breathing (10:15-min) for 8 weeks. The stepping reaction time will be assessed by the choice stepping reaction time (CSRT). The Balance will be determined using a Time up and Go test (TUG) an d Berg balance scale (BBS). All the outcomes will be examined at baseline, and 8 weeks of the intervention.

ELIGIBILITY:
Inclusion Criteria:

* All participants with a history of COPD
* Adults ranging from 55- 70 years old of both genders.
* Medically stable

Exclusion Criteria:

* Obesity (BMI ≥ 30 kg/m2)
* History of Pneumonia
* Diaphragmatic hernia, clinical evidence of phrenic nerve injury, recent abdominal or thoracic surgery, or history of traumatic lesion possibly affecting diaphragm.
* History of Myocardial infarction and/or cardiothoracic surgery
* orthopedics, or neurological that may interfere the intervention.
* Visual impairments, vestibular disorders, and postural hypotension.
* Dementia that interferes with the ability to follow instructions.

Ages: 55 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2024-08-22 (Actual); Primary Completion 2025-08-15 (Estimated); Study Completion 2025-11-15 (Estimated)

PRIMARY OUTCOMES:
stepping reaction time | up to 8 weeks
  stepping reaction time will be assessed by choice stepping reaction time test. The test procedure is as follows: when the stepping target is illuminated in a random order, the subject steps onto the illuminated target as quickly as possible.4 The faster the reaction, the shorter the reaction time.
Balance | up to 8 weeks
  Balance Balance will be assessed by berg balance scale, the balance score ranges from 0 to 56, with lower scores indicating increased risk of balance loss and higher scores indicating improved functional mobility. Time up and go test (TUG)n Score < 10 seconds = normal < 20 seconds = good mobility; can walk outside alone; does not require a walking aid < 30 seconds = walking and balance problems; cannot walk outside alone; requires walking aid.

CONTACTS AND LOCATIONS:
Overall Officials: Mohammed S Saif, Ph.D, Study Director — National institute for Gerontology
Locations (1):
- Kz Hospital, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: No